CLINICAL TRIAL: NCT05993416
Title: Treatment of Primary Hyperoxaluria Type 1 With Nedosiran
Status: No longer available | Type: Expanded Access
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Other Study IDs: DCR-PHXC-401
Record Dates: First submitted 2023-08-06; First posted 2023-08-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1)
MeSH Terms: conditions — Primary hyperoxaluria type 1 | interventions — nedosiran

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Nedosiran — In adults and in adolescents (aged 12-17 years) weighing greater than or equal to (>=) 50 kilograms (kg), Nedosiran will be administered via subcutaneous (SC) injection once monthly at a dose of 170 milligrams (mg). In adults and adolescents weighing < 50 kg, nedosiran will be administered once monthly at a dose of 136 mg. The dose for participants aged 6 to 11 years will be 3.5 mg/kg monthly, not to exceed 170 mg.

SUMMARY:
The purpose of this program is to provide participants with access to an investigational drug, nedosiran, for treatment of primary hyperoxaluria type 1 (PH1). Eligible participants may receive nedosiran in this program until the drug is commercially available or until Novo Nordisk terminates the program, whichever comes first. Novo Nordisk may terminate the program at any time for any reason, including if the drug receives regulatory approval and becomes commercially available, or if the drug does not receive regulatory approval. Nedosiran will be given once a month with a thin needle in the thigh or abdomen. The study doctor will ask the participant to come to the clinic monthly. The study doctor may allow participant to take nedosiran at home for self-administration. The participant should let the doctor know if they are unable to make a visit so it can be rescheduled. Participants to inform the study doctor of any medications they are taking, including over the counter medicines, vitamins, and herbal medicines. If any medications change in dose, or new medications are added, participants should inform the study doctor. Study doctor should be informed of any new or continued health problems or any changes in the participant's health.

ELIGIBILITY:
Early Access Eligibility Criteria:

* Written, signed, and dated informed patient/parent consent; and for patients who were minors, age-appropriate assent (performed according to local regulations)
* Male or female patients at least 2 years of age
* Genetically-confirmed diagnosis of PH1
* Accessible for treatment and follow-up and be able to comply with treatment monitoring requirements
* Not eligible for an ongoing RNAi therapy trial and not participating simultaneously in any interventional clinical research study
* Patients with PH1 that are not satisfactorily treated with current standard of care; i.e., 24-hour urinary oxalate (Uox) excretion ≥ 0.7 (millimoles) mmol for participants 18 years and older, or greater or lesser than (≥) 0.7 mmol per 1.73 metre square (m^2) body surface area (BSA) for participants less than 18 years of age
* Estimated GFR at screening ≥ 30 millilitres per minute (mL/min) normalized to 1.73 m^2 BSA
* No renal or hepatic transplantation; prior or planned within the treatment period
* No documented evidence of clinical manifestations of systemic oxalosis (including pre existing retinal, heart, or skin calcifications, or history of severe bone pain, pathological fractures, or bone deformations)
* Patient not currently on dialysis
* Plasma oxalate ≤ 30 micromoles per litre (μmol/L)
* Female patients not breastfeeding or pregnant
* The potential benefit for the individual patient justifies the potential risks of treatment as per prescribing physician judgment

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult